CLINICAL TRIAL: NCT02510404
Title: Treatment of EBV, CMV, and Adenovirus Infections in Primary Immunodeficiency Disorders With Viral-specific Cytotoxic T-Lymphocytes
Brief Title: Multivirus-specific Cytotoxic T Lymphocytes (mCTL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catherine Bollard (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Sponsor-Investigator, Catherine Bollard, Director- Program for Cell Enhancement and Technologies for Immunotherapy (CETI), Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TREPID
Record Dates: First submitted 2015-07-13; First posted 2015-07-29 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Refractory Viral Infections
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mCTLs against three viruss (Experimental): The investigator will use 3 different dose levels starting with 5 x 106 (a T cell number more than an order of magnitude lower than that administered at the time of an unmanipulated marrow infusion), followed by 1 x 107 and a final dose 2 x 107 mCTLs/m2. They will give the option of administering 2 additional doses (at the same level) of the same or different cell lines, 28 days after the first dose, in subjects that have limited or no improvement in viral count after one dose in the absence of any toxicities attributable to the infusion,or who receive other therapy that may affect the persistence or function of the infused mCTLs.
  Interventions: Biological: mCTLs

INTERVENTIONS:
Biological: mCTLs — The investigators have elected to limit this phase I study to PIDD patients with active viral infections unable to be controlled with standard pharmacotherapy, who are therefore likely to benefit from mCTLs treatment. This trial will be performed as dose-escalation study. Patients will be evaluated for matched lines from a bank of third-party mCTLs, derived from CMV seropositive donors. These lines will have been used clinically in prior clinical trials, with safety demonstrated in the post-HSCT setting.

SUMMARY:
PIDD represent an expanding group of genetic disorders that compromise immunity against bacteria, viruses, and fungi. The most severe forms of PIDD cause profound susceptibility to opportunistic infections due to impaired or absent T-cell immunity. These diseases can be rapidly fatal unless treated via hematopoietic stem cell transplantation (HSCT). Chronic viral illnesses are a common presenting feature of many of these disorders, and studies have shown that survival of HSCT is profoundly impacted by the patient's pre-transplant disease status. Primary infections with viruses such as cytomegalovirus (CMV) and Epstein-Barr virus (EBV) are common, and respiratory viruses such as adenovirus also frequently cause infection. In patients with severe combined immunodeficiency (SCID), a prior study identified these viruses as the most common causes of mortality in the immediate period following HSCT. Though some forms of PIDD are amenable to HSCT without requiring conditioning chemotherapy, many forms require a variable degree of pre-conditioning to ensure that stable engraftment of the donor cells is achieved. The administration of cytotoxic chemotherapy used in the conditioning regimens can however increase the risk for regimen related toxicity and for some patients (especially those with active viral infections) this risk is particularly high, leading to high treatment related mortality rates. For these reasons, many such patients are not even considered candidates for HSCT or are delayed getting to HSCT and ultimately succumb to infection before they can receive the transplant.

The primary objective of this study is to determine the safety of administering third-party multivirus-specific cytotoxic T lymphocytes (mCTL) from adult CMV seropositive donors to treat refractory viral infections in patients with primary immunodeficiency disorders (PIDD) prior to hematopoietic stem cell transplantation (HSCT).

DETAILED DESCRIPTION:
Since recovery of virus-specific T cells is clearly associated with protection from infection with each of these viruses, adoptive immunotherapy to decrease the time to immune reconstitution is an attractive approach. Virus-specific T cells generated by repeated stimulation with antigen presenting cells (APCs) expressing viral antigens have been evaluated in clinical trials to prevent and treat viral infections in immunocompromised hosts. This approach eliminates alloreactive T cells.

To broaden the specificity of single CTL lines to include the three most common viral pathogens of stem cell recipients, investigators reactivated CMV and adenovirus-specific T cells by using mononuclear cells transduced with a recombinant adenoviral vector encoding the CMV antigen pp65 (Ad5f35CMVpp65). Subsequent stimulations with EBV-LCL transduced with the same vector both reactivated EBV-specific T cells and maintained the expansion of the activated adenovirus and CMV-specific T cells. This method reliably produced CTLs with cytotoxic function specific for all three viruses, which investigators infused into 14 stem cell recipients in a Phase I prophylaxis study. They observed recovery of immunity to CMV and EBV in all patients but an increase in adenovirus-specific T cells was only seen in patients who had evidence of adenovirus infection pre-infusion. A follow-up study in which the frequency of adenovirus-specific T cells was increased in the infused CTLs produced similar results, thus highlighting the importance of endogenous antigen to promote the expansion of infused T cells in vivo. Nevertheless, all patients in both clinical trials with pre-infusion CMV, adenovirus or EBV infection or reactivation were able to clear the infection, including one patient with severe adenoviral pneumonia requiring ventilatory support. CTLs recognizing multiple antigens can therefore produce clinically relevant effects against all three viruses.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of primary immunodeficiency with established plan to undergo myeloablative or non-myeloablative allogeneic hematopoietic stem cell transplant for treatment thereof or diagnosis of a form of primary immunodeficiency for which hematopoietic stem cell transplantation is not indicated.
2. Active infection with EBV, CMV, and/or Adenovirus, unable to be successfully controlled with standard therapy.
3. Steroids less than 0.5 mg/kg/day prednisone
4. Karnofsky/Lansky score of ≥ 50
5. ANC greater than 500/µL.
6. Bilirubin <2x, AST <3x, Serum creatinine <2x upper limit of normal, Hgb >8.0
7. Pulse oximetry of > 90% on room air
8. Negative pregnancy test (if female of childbearing potential)
9. Patient or parent/guardian capable of providing informed consent.

Exclusion Criteria:

1. Patients with other uncontrolled infections (see 2.3.2 for definitions)
2. Patients who received ATG, Campath, or other T cell immunosuppressive monoclonal antibodies in the last 28 days
3. Received donor lymphocyte infusion in last 28 days
4. Diagnosis of Omenn's syndrome or MHC class I deficiency
5. Active and uncontrolled malignancy
6. Pregnant or lactating
7. Unable to wean steroids to ≤0.5 mg/kg/day prednisone.
8. Patients with Grade 3 hyperbilirubinemia

Ages: 4 Weeks to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-06-08 (Actual)

PRIMARY OUTCOMES:
Assessments of patients with adverse events after mCTLs infusion | 45 days
  The safety endpoint will be defined as acute GvHD grades III-IV related to the T cell product within 45 days of the last VST dose and that are not due to the pre-existing infection or the original malignancy or pre-existing co-morbidities as defined by the NCI Common Terminology Criteria for Adverse Events (CTCAE)

SECONDARY OUTCOMES:
Assessments of viral load response to the mCTLs infusion | 12 months
  Increase in viral load of at least 50% from baseline or dissemination to other sites of disease.
Assessments of Antiviral Immunity | 12 months
  Patient serum and peripheral blood mononuclear cells will be monitored for virus-specific activity by phenotypic and functional studies including ELIspot with appropriate viral specific peptide mixtures and available HLA-restricted epitope peptides, intracellular cytokine staining, serum cytokine profiling and/or other assays as they become available for immune profiling purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Bollard, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Childrens National Medical Center, Washington D.C., District of Columbia, United States